CLINICAL TRIAL: NCT03290599
Title: Effect of Preoperative Hospitalization Duration on Post-operative Cognitive Dysfunction in Patients Who Underwent Hip Surgery Under Regional Anesthesia
Brief Title: Effect of Preoperative Hospitalization Duration on Post-operative Cognitive Dysfunction
Status: Completed | Type: Observational
Sponsor: Burcu Ozalp Horsanali (Other)
Responsible Party: Sponsor-Investigator, Burcu Ozalp Horsanali, Burcu OZALP HORSANALI, Kackar State Hospital
Organization: Kackar State Hospital (Other)
Other Study IDs: 1
Record Dates: First submitted 2017-09-17; First posted 2017-09-25 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Post Operative Cognitive Dysfunction
Keywords: Cognitive dysfunction; Hip Surgery; Mini mental Test,; Preoperative Hospitalisation; Spinal Anesthesia
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No Post operative cognitive dysfunction: Patients who did not have any change or a change less than 4 points between MMT1 and MMT3
  Interventions: Other: Mini Mental and Modified Mini Mental Test
- Post operative cognitive dysfunction: Patients with a difference more than 4 points between MMT1 and MMT3
  Interventions: Other: Mini Mental and Modified Mini Mental Test

INTERVENTIONS:
Other: Mini Mental and Modified Mini Mental Test — Mini Mental Test was used for literate patients and Modified mini mental test was used for illiterated patients

SUMMARY:
Post-operative cognitive dysfunction is defined as a decrease in cognitive functions which develop following surgery and anesthesia administration that can last up to weeks or even months after surgery. In this study, our main objective was to investigate the effect of preoperative hospitalisation period on early post operative cognitive dysfunction development and its risk factors in patients who underwent total hip replacement surgery for hip fractures under regional anesthesia.

DETAILED DESCRIPTION:
The study evaluated Mini Mental Test scores of patients who received total hip replacement surgery in Izmir Bozyaka Training and Research Hospital from November 2013 to September 2014. In the assessment, Mini Mental Test (MMT) was used for literate and Modified Mini Mental Test (MMMT) was used for illiterate patients. Test scores were obtained on the initial admission day (MMT1), 24 hours prior to surgery (MMT2) and 24 hours after the surgery (MMT3). A drop of 4 points or more between each test was defined as significant cognitive dysfunction development. Patients who did not have any change or a change less than 4 points between MMT1 and MMT3 were grouped as "no cognitive dysfunction" (Group 1) and patients with a difference more than 4 points between MMT1 and MMT3 were grouped as "cognitive dysfunction" (Group 2). All analyses were performed using those 2 patient groups.

Patients who were planned to undergo total hip replacement surgery without cement over 18 years of age and within ASA Group 1, 2 and 3 according to ASA physical status score were included in the study.

Patients younger than 18, who did not speak Turkish, with known cancer history, previous steroid treatment, SVO history in last 6 months, with central nervous system diseases (current meningitis, encephalitis, tumors, major degenerative diseases), with dementia, Alzheimer's and Parkinson's Disease, pregnant patients, patients with neuropsychiatric diseases or received antidepressant, antipsychotic or anticonvulsive treatment in the last 6 months, uncooperative patients, patients with substance abuse problems, patients with severe organ failure (end-stage liver failure, dialysis-dependent kidney failure), patients who required ICU following surgery, patients where regional anesthesia was contraindicated (Idiopathic intracranial hypertension (IIH), clotting disorders, infection on operational site) were excluded from the study.

No premedication was done on patients during preoperative period. Hydration during preoperative period was done by IV 0.9% NaCl aqueous solution with a fasting period of 6-10 hours prior to surgery.

In our study, combined spinal-epidural anesthesia was used for anesthesia for all the patients. Surgical intervention was allowed on the patients with sensory block on T8 dermatome levels. Patients also received 0.5 mg IV bolus midazolam with Ramsey Sedation Scale 3.

During anesthesia, systolic blood pressure decreases more than 20% compared to preoperative period was defined as hypotension. 5 mg IV Ephedrine was administered to the patients when their arterial blood pressure levels stayed 50mmHg and below despite fluid replacement. Bradycardia was defined as pulses below 40 bpm and was treated with 0.5 mg IV atropine.

Postoperative pain management was planned according to Visual Analogue Scale (VAS). In patients with VAS score 3 and above, 10 ml isobaric bupivacaine 0.125% was administered through epidural catheter. No additional medication (opiates or NSAIDs) were used for analgesia.

Demographics, education levels, employment status, operation indications, ASA scores, comorbid diseases and tobacco use of all patients were questioned and recorded. Scores of MMT or MMMT of patients on their initial admission, 24 hours prior to surgery and 24 hours after surgery and its parameters were all recorded and grouped.

The period from the initial admission to the surgery date was calculated and recorded. Patients' hemoglobin, hematocrit, serum electrolyte levels on their admission, preoperative and postoperative periods were recorded.

Finally, anesthesia duration, surgery duration, administered midazolam, atropine and ephedrine doses, crystalloid, colloid, blood and blood products used during surgery and total blood loss volume were all recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were planned to undergo total hip replacement surgery without cement over 18 years of age and within ASA Group 1, 2 and 3 according to ASA physical status score were included in the study.

Exclusion Criteria:

* Patients younger than 18, who did not speak Turkish, with known cancer history, previous steroid treatment, SVO history in last 6 months, with central nervous system diseases (current meningitis, encephalitis, tumors, major degenerative diseases), with dementia, Alzheimer's and Parkinson's Disease, pregnant patients, patients with neuropsychiatric diseases or received antidepressant, antipsychotic or anticonvulsive treatment in the last 6 months, uncooperative patients, patients with substance abuse problems, patients with severe organ failure (end-stage liver failure, dialysis-dependent kidney failure), patients who required ICU following surgery, patients where regional anesthesia was contraindicated (Idiopathic intracranial hypertension (IIH), clotting disorders, infection on operational site) were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who underwent total hip replacement surgery over 18 aged
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2013-11-01 (Actual); Primary Completion 2014-09-30 (Actual); Study Completion 2014-09-30 (Actual)

PRIMARY OUTCOMES:
Post operative Cognitive Dysfunction | change of Mini mental test score from hospitalisation time to post operative 24th hour
  Mini mental test

IPD SHARING:
Plan to Share IPD: No